CLINICAL TRIAL: NCT06609499
Title: Standard Gum Elastic Bougie Versus Flexible-tip Bougie: Evaluation of Airway Adjuncts for Intubation in Entrapped Patients With Difficult Airway Access - a Randomised, Controlled Trial
Brief Title: Evaluation of Airway Adjuncts for Intubation in Entrapped Patients With Difficult Airway Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uniwersytet Radomski im. Kazimierza Pułaskiego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 04/2024
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Airway Obstruction
Keywords: tracheal intubation; trauma; entrapped patients,; introducer; flexible-tip bougie
MeSH Terms: conditions — Airway Obstruction; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Masking Description: A single digit number will be allocated to each of the two studied devices i.e. 1 for the flexible-tip bougie and 2 for the standard gum elastic bougie. Each study participant will be asked to randomly give a number (either 1 or 2) and will then be given the corresponding tracheal tube introducer to use. The maximum number of intubation attempts is limited to three per device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flexible-tip Bougie Group (Experimental): Paramedics using the flexible-tip bougie (the STIG)
  Interventions: Device: Flexible-tip Bougie
- Gum-elastic bougie Group (Active Comparator): Paramedics using the gum-elastic bougie
  Interventions: Device: Gum-elastic Bougie

INTERVENTIONS:
Device: Flexible-tip Bougie — The device is used for intubation and then the manikin is ventilated
  Arms: Flexible-tip Bougie Group
Device: Gum-elastic Bougie — The device is used for intubation and then the manikin is ventilated
  Arms: Gum-elastic bougie Group

SUMMARY:
The aim of this clinical trial is to evaluate two airway adjuncts for intubation in a simulated condition of an entrapped trauma patient with simultaneous cervical spine immobilisation. All the studied devices are evaluated by fully-qualified and experienced paramedics (both male and female). The main questions it aims to answer are:

Which device requires the shortest time required to achieve a successful intubation and ventilation? What is the first attempt success rate of the studied devices? Which device is the easiest to use and the most user-friendly? Study participants will evaluate two different airway adjuncts for intubation in a restricted access to the entrapped trauma patient's airway. The maximum number of insertion attempts is limited to three per device.

DETAILED DESCRIPTION:
A written informed consent will be obtained from all study participants. Only qualified paramedics will participate in the study. Their experience varies between four and eight years of practice after completion of paramedic training. All study participants had never used the flexible-tip bougie but had a routine intubation experience with the standard gum elastic bougie (more than 40 intubations previously performed).

A 10-minute lecture will be delivered before the start of the study. It will explain how to use the STIG. Following the lecture all participants will be able to familiarise themselves with the equipment and practice for 30 minutes. A skill station will be set up containing an intubation manikin AT Kelly Torso (Laerdal Medical AS, Stavanger, Norway). A reduced movement of the cervical spine will be achieved by application of a Patriot® cervical collar (Össur hf., Reykjavik, Iceland). After completion of the initial practice the intubation manikin with the cervical collar on wall be placed on and secured to the driver's seat of a FIAT Bravo car (FIAT S.p.A., Turin, Italy). The car will then be positioned on its left side and secured in place by firemen from a local fire brigade. The access to the manikin will only allowed from the front i.e. through the opening created after removal of the windscreen. A single digit number will be allocated to each of the two studied devices i.e. 1 for the flexible-tip bougie and 2 for the standard gum elastic bougie (SUMI Sp. z o.o., Sp. K., Sulejówek, Poland). Each study participant will be asked to randomly give a number (either 1 or 2) and will then be given the corresponding tracheal tube introducer to use. The maximum number of intubation attempts is limited to three per device. The time required to intubate and successfully ventilate (Ti) the manikin will be recorded. It will be measured using a stopwatch of a mobile phone (Apple Inc., Cupertino, California, USA). Efficacy of intubation and the ease of use by the operator will also be assessed. The latter will be measured using an 11-point numerical rating scale (NRS) where 0 corresponds to a very difficult to use device and 10 indicates an easy to use and user-friendly introducer. Size 7.5 tracheal tube (SUMI Sp. z o.o., Sp. K., Sulejówek, Poland) will be utilised in the study. A manual resuscitator (Ambu A/S, Ballerup, Denmark) will be used for ventilation and will be readily available to the paramedics. The standard Macintosh-blade laryngoscope (New Waseem Trading Co., Sialkot, Pakistan) will be utilised for direct laryngoscopy. Size three blade will be used. The study participants will perform all intubations with each of the two tracheal tube introducers. A failed intubation will be defined as an attempt during which the trachea cannot be intubated or an attempt that lasts longer than 120 seconds. Only those who failed to intubate will be allowed another attempt. All the obtained data will be analysed using Microsoft Office Excel 2021 spreadsheet (Microsoft Corporation, Redmond, WA, USA) and GraphPad Prism (GraphPad Software, Boston, MA, USA). The Kolmogorov-Smirnov test will be utilised to determine whether the analysed variables matches the characteristics of a normal distribution. A paired Student t-test and the Wilcoxon signed-rank test will be used for data analysis. Based on our previous unpublished pilot study and assuming that the overall success rate of intubation in patients with a difficult airway will be 90% (α =0.05, 2-sided, β =0.1), 46 participants are required. The final adjusted sample size, allowing a drop-out rate of about 10%, will be 50 and this is the final number of participants enrolled into the study. A p value of less than 0.05 (p<0.05) is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* fully-qualified paramedics
* at least four years of practice after finishing paramedic training
* active (working) paramedics

Exclusion Criteria:

* paramedics in training
* retired paramedics
* lack of written informed consent

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Successful intubation time | From the date of randomization until the date of documented completion, assessed up to four months
  The time required to intubate and successfully ventilate the manikin

SECONDARY OUTCOMES:
First attempt success rate of intubation | From the date of randomization until the date of documented completion, assessed up to four months
  The efficacy of evaluated airway adjuncts
The ease of use and user-friendliness | From the date of randomization until the date of documented completion, assessed up to four months
  Device evaluation using the numerical rating scale (NRS). It is an 11-point scale where 0 corresponds to a very difficult to use device and 10 indicates an easy to use and user-friendly device.

CONTACTS AND LOCATIONS:
Overall Officials: Dawid J Aleksandrowicz, PhD, Principal Investigator — University of Radom
Locations (1):
- University of Radom, Radom, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No